CLINICAL TRIAL: NCT07337486
Title: "Evaluation of a Non-Pharmacological Skin Care Intervention for the Prevention and Treatment of Skin Toxicities Caused by Immunotherapy in Cancer Patients"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IIBSP-CUT-2021-109
Record Dates: First submitted 2024-06-21; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2024-06

CONDITIONS: Skin Toxicity in Patients on Checkpoint Inhibitors
Keywords: Immunotherapy; immune-mediated skin toxicity; Prevention; Checkpoint-inhibitors; Skin hygiene and hydration care; Cancer; Immuno-mediated cutaneous toxicity (pruritus and/or xerosis) in patients undergoing immunotherapy for cancer
MeSH Terms: conditions — Neoplasms | interventions — Niacinamide; argan oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Niacinamide and Shea Butter (Experimental)
  Interventions: Other: Shea Butter and Niacinamide
- Argan Oil and Coconut Butter (Active Comparator)
  Interventions: Other: Argan Oil and Coconut Butter

INTERVENTIONS:
Other: Shea Butter and Niacinamide — Thus, this study seeks to contribute novel insights into managing patients undergoing active immunotherapy, a field that remains relatively unexplored. Dermocosmetic products used in both armes of this trial are already approved for over-the-counter use, ensuring accessibility without prescription.
  Arms: Niacinamide and Shea Butter
Other: Argan Oil and Coconut Butter — Thus, this study seeks to contribute novel insights into managing patients undergoing active immunotherapy, a field that remains relatively unexplored. Dermocosmetic products used in both armes of this trial are already approved for over-the-counter use, ensuring accessibility without prescription.
  Arms: Argan Oil and Coconut Butter

SUMMARY:
Due to recent approvals, a significant number of adult cancer patients are undergoing treatment with checkpoint inhibitor antibodies. While these treatments have revolutionized cancer care, they come with inherent risks of toxicities, primarily mediated by the patient's own immune system.

Among the most common side effects are dermatological toxicities, which although generally mild, significantly impact patients' quality of life. These issues are often underdiagnosed and lack proactive interventions. This study aims to demonstrate that proactive measures using Niacinamide and Shea Butter can either prevent or mitigate the severity of these toxicities.

Thus, this study seeks to contribute novel insights into managing patients undergoing active immunotherapy, a field that remains relatively unexplored. Dermocosmetic products used in both armes of this trial are already approved for over-the-counter use, ensuring accessibility without prescription.

Study Hypothesis: The prophylactic use of Niacinamide and Shea Butter in dermocosmetic products reduces the frequency and severity of immune-mediated skin toxicities in cancer patients receiving checkpoint inhibitor antibodies.

This single-center trial will be conducted at Hospital de la Santa Creu i Sant Pau, employing a parallel arm design with randomization overseen by the center's statistician. Participants will be randomly assigned to either arm, with an active control group to monitor dermocosmetic product usage frequency and type. The blinding protocol will be single-blind to ensure unbiased evaluation.

The study aims to assess the incidence of pruritus among adult cancer patients receiving checkpoint inhibitor antibodies, correlating these findings with the efficacy of dermocosmetic products containing Niacinamide and Shea Butter. Additionally, it will evaluate the impact on the quality of life of these patients.

The intervention group will receive soap and an emollient formulated with Shea Butter and Niacinamide, while the control group will use products containing Argan Oil and Coconut Butter. Both groups will undergo a 6-month treatment regimen.

Key endpoints include:

* Skin pruritus
* Relationship between skin condition and quality of life Consecutive non-probabilistic sampling will be used to recruit all patients with solid tumors initiating immunotherapy.

Using GranMo calculator version 7.2 with 95% confidence and a precision of +/- 0.07, the study calculated a sample size of 128 patients. Recruitment will aim for 130 patients to account for potential attrition, split evenly between Arm 1 and Arm 2.

Data analysis will involve importing, cleaning, and recoding variables followed by univariate analysis using IBM SPSS v.25 The study will adhere strictly to international ethical standards for clinical research, including the Declaration of Helsinki and Good Clinical Practice guidelines. Participants will be fully informed about the study's nature, objectives, procedures, potential risks, benefits, and their right to withdraw without impact on their care.

An information/consent form has been designed accordingly. Participants will receive hygiene and hydration products at no cost, though no financial compensation will be provided.

Monitoring, auditing, reviews by the CEIC, and regulatory inspections will be conducted to ensure adherence to protocol and regulatory requirements.

The choice of control treatment aims to replicate real-world conditions while assessing approved products. Participants will be followed for 6 months from informed consent signing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Diagnosed with any solid cancer
* Initiating treatment with checkpoint inhibitor antibodies
* Able to speak and understand Spanish and/or Catalan

Exclusion Criteria:

* Unable to sign informed consent
* Unable to comprehend the study for giving consent
* Language barrier: Does not speak or understand Spanish or Catalan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Objective 1: Itching | 19 months
  Evaluate the occurrence of itching in adult cancer patients receiving treatment with Checkpoint Inhibitor Antibodies in relation to prevention with the use of dermocosmetic products based on Niacinamide and Shea Butter. The itch is measured using the itch intensity scale. It is a scale validated in both English and Spanish.
Objective 2: Skin quality of life | 19 months
  Evaluate the quality of life of adult cancer patients receiving treatment with Checkpoint Inhibitor Antibodies regarding skin health. The quality of life related to skin is evaluated using the Dermatology Life Quality Index (DLQI).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martins F, Sofiya L, Sykiotis GP, Lamine F, Maillard M, Fraga M, Shabafrouz K, Ribi C, Cairoli A, Guex-Crosier Y, Kuntzer T, Michielin O, Peters S, Coukos G, Spertini F, Thompson JA, Obeid M. Adverse effects of immune-checkpoint inhibitors: epidemiology, management and surveillance. Nat Rev Clin Oncol. 2019 Sep;16(9):563-580. doi: 10.1038/s41571-019-0218-0. PMID 31092901
- [Result] Davies M. How Checkpoint Inhibitors Are Changing the Treatment Paradigm in Solid Tumors: What Advanced Practitioners in Oncology Need to Know. J Adv Pract Oncol. 2016 Jul-Aug;7(5):498-509. Epub 2016 Jul 1. PMID 29282426
- [Result] Belum VR, Benhuri B, Postow MA, Hellmann MD, Lesokhin AM, Segal NH, Motzer RJ, Wu S, Busam KJ, Wolchok JD, Lacouture ME. Characterisation and management of dermatologic adverse events to agents targeting the PD-1 receptor. Eur J Cancer. 2016 Jun;60:12-25. doi: 10.1016/j.ejca.2016.02.010. Epub 2016 Apr 1. PMID 27043866
- [Result] Haanen JBAG, Carbonnel F, Robert C, Kerr KM, Peters S, Larkin J, Jordan K; ESMO Guidelines Committee. Management of toxicities from immunotherapy: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv119-iv142. doi: 10.1093/annonc/mdx225. No abstract available. PMID 28881921
- [Result] Sibaud V. Dermatologic Reactions to Immune Checkpoint Inhibitors : Skin Toxicities and Immunotherapy. Am J Clin Dermatol. 2018 Jun;19(3):345-361. doi: 10.1007/s40257-017-0336-3. PMID 29256113
- [Result] Lacouture M, Sibaud V. Toxic Side Effects of Targeted Therapies and Immunotherapies Affecting the Skin, Oral Mucosa, Hair, and Nails. Am J Clin Dermatol. 2018 Nov;19(Suppl 1):31-39. doi: 10.1007/s40257-018-0384-3. PMID 30374901
- [Result] Macdonald JB, Macdonald B, Golitz LE, LoRusso P, Sekulic A. Cutaneous adverse effects of targeted therapies: Part I: Inhibitors of the cellular membrane. J Am Acad Dermatol. 2015 Feb;72(2):203-18; quiz 219-20. doi: 10.1016/j.jaad.2014.07.032. PMID 25592338
- [Result] Anforth R, Fernandez-Penas P, Long GV. Cutaneous toxicities of RAF inhibitors. Lancet Oncol. 2013 Jan;14(1):e11-8. doi: 10.1016/S1470-2045(12)70413-8. PMID 23276366